CLINICAL TRIAL: NCT01269619
Title: Comparative Study of Static and Dynamic Back Supports for Lower Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Yigal Bronstein, M.D., Wolfson Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUG-001
Record Dates: First submitted 2011-01-02; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-12

CONDITIONS: Low Back Pain, Mechanical
Keywords: back pain; posture; lumbar support; dynamic support
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dynamic (Experimental): Use of Dynamic back support
  Interventions: Device: Dynamic back support
- Static (Active Comparator): Use of static back support
  Interventions: Device: Static back support

INTERVENTIONS:
Device: Dynamic back support — A dynamic back support which provides pressure on the lumbar without pressure on the abdomen
  Other Names: hug by Koala
  Arms: Dynamic
Device: Static back support — A standard wrap-around sacro lumbar support
  Other Names: Oppo sacro lumbar support
  Arms: Static

SUMMARY:
Lower back pain is one of the most common conditions affecting humans. Lower back supports are a common device used in order to alleviate the pain. All the available back supports are wrapped around the lower back and abdomen and act as static support devices. "The hug" is a new dynamic back support where the participant actively improves his/her posture and strengthens the muscle of the lower back. This trial compares both devices and their effect on reducing lower back pain.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent back pain
* use analgesics

Exclusion Criteria:

* Pregnant women
* malignancy
* infection
* neurological condition
* surgical candidate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Reduction in back pain | 3 weeks

SECONDARY OUTCOMES:
Patient satisfaction | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Medical Center, Holon, Israel